CLINICAL TRIAL: NCT01811329
Title: Effects of Dairy Fat on Postprandial Inflammation- Phase 1
Brief Title: Determine How Consumption of Dairy Fat Fractions Rich in Phospholipids and Proteins Influence Inflammation in the Fed State-Phase 1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 264297-1; 264297-1 (Other: UC Davis IRB)
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Palm fat (Active Comparator): The amount of calories in the shake will be equivalent to 30% of each participant's calculated energy expenditure. The macronutrient composition of the shake as a percent of energy will be: 45% fat, 40% carbohydrate and 15% protein. The shake will contain palm fat, frozen fruit, glucose polymer, and protein powder.
  Interventions: Dietary Supplement: Palm fat
- Palm fat + MFGM (Experimental): The amount of calories in the shake will be equivalent to 30% of each participant's calculated energy expenditure. The macronutrient composition of the shake as a percent of energy will be: 45% fat, 40% carbohydrate and 15% protein. The shake will contain palm fat, frozen fruit, glucose polymer, and BPC50, a dairy fraction rich in milk fat globule membrane proteins and phospholipids. Fifty percent of the shake's fat will be derived from BPC50.
  Interventions: Dietary Supplement: Palm fat + MFGM
- Dairy fat (Active Comparator): The amount of calories in the shake will be equivalent to 30% of each participant's calculated energy expenditure. The macronutrient composition of the shake as a percent of energy will be: 45% fat, 40% carbohydrate and 15% protein. The shake will contain whipping cream, frozen fruit, glucose polymer, and protein powder.
  Interventions: Dietary Supplement: Dairy fat
- Dairy fat + MFGM (Experimental): The amount of calories in the shake will be equivalent to 30% of each participant's calculated energy expenditure. The macronutrient composition of the shake as a percent of energy will be: 45% fat, 40% carbohydrate and 15% protein. The shake will contain whipping cream, frozen fruit, glucose polymer, and BPC50, a dairy fraction rich in milk fat globule membrane proteins and phospholipids. Fifty percent of the shake's fat will be derived from BPC50.
  Interventions: Dietary Supplement: Dairy fat + MFGM

INTERVENTIONS:
Dietary Supplement: Dairy fat
  Arms: Dairy fat
Dietary Supplement: Dairy fat + MFGM — BPC50, a dairy fraction rich in milk fat globule membrane proteins and phospholipids manufactured by Fonterra, will make up 50% of the shake's total fat.
  Arms: Dairy fat + MFGM
Dietary Supplement: Palm fat
  Arms: Palm fat
Dietary Supplement: Palm fat + MFGM — BPC50, a dairy fraction rich in milk fat globule membrane proteins and phospholipids manufactured by Fonterra, will make up 50% of the shake's total fat.
  Arms: Palm fat + MFGM

SUMMARY:
Phase 1 of this study involves determining how consumption of dairy fat fractions rich in milk fat globule membrane influences postprandial inflammation in participants with metabolic syndrome or obesity during a high dietary fat challenge in a six-hour period.

DETAILED DESCRIPTION:
Phase 1 is a randomized crossover study designed to determine how inclusion of dairy fractions rich in milk fat globule membrane (MFGM) to shakes rich in dairy or palm fat influence postprandial inflammation. Participants who have 2 or more risk factors of metabolic syndrome or BMI ≥ 30 will consume four shakes on separate days. The four shakes are: high dairy fat, high dairy fat + MFGM, high palm fat, high palm fat + MFGM.

Eligible participants will arrive to the Western Human Nutrition Research Center (WHNRC) at the University of California (UC) Davis campus on the morning of each test day after a 10-12-hr overnight fast. Upon arrival participants will fill out a questionnaire about their dietary and medication intakes and physical activity for the past 72 hours to ensure compliance. Compliant participants' weight and blood pressure will be measured and a fasting blood draw will be taken before participants consume their test meal. Participants will only consume this test meal and water freely for the duration of the test day. Blood will be drawn serially at 1, 3 and 6 hours postprandially. Participants will be tested on the additional three arms on three different spaced apart by two weeks.

On the third or fourth test day, participants' body composition and bone mineral density will be measured by dual x-ray absorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Two or more components of metabolic syndrome:

Central obesity (waist circumference greater than 40 inches for men and 35 inches for women); fasting blood triglycerides greater than or equal to 150 mg/dL; plasma HDL cholesterol (Less than 40 mg/dL for men and less than 50 mg/dL for women); blood pressure greater than or equal to 130/85 mmHg; fasting glucose greater than or equal to 100 mg/dL

or

- BMI equal to or greater than 30

Exclusion Criteria:

Metabolic Disorders:

* BMI > 40
* Body weight more than 400 lbs.
* Any immune related diseases such as autoimmune disease, rheumatoid arthritis, asthma,
* Gastrointestinal disorders including Crohn's Disease, colitis, diverticulitis, irritable bowel disease, celiac, malabsorption syndrome
* Cancer
* Known presence of significant metabolic disease which could impact the results of the study (i.e. hepatic, renal disease)
* Type II diabetes
* Use of over-the-counter anti-obesity agents (e.g. containing phenylpropanolamine, ephedrine, and/or caffeine) within the last 12 weeks
* Use of corticoid steroids within the last 12 weeks
* Daily use of anti-inflammatory pain medication
* Self report of eating disorder
* Poor vein assessment determined by WHNRC's phlebotomist

Dietary/supplements:

* Known allergy or intolerance to study food (lactose intolerance, dairy, wheat allergies)
* Vegetarian (defined as abstinence from consumption of eggs, dairy, poultry, beef and pork)
* More than 1 serving of fish per week
* More than 14 grams of fiber per 1000 kcal per day
* Less than 16:1 of total dietary omega 6: Omega 3 ratio
* More than 1% of daily energy as trans fats
* Initiation of anti-inflammatory supplemental fish, krill, flax, borage and primrose seed oils within the last 12 weeks
* Dietary supplements consisting of concentrated soy isoflavones, resveratrol, other polyphenols identified as modulators of inflammation Medications
* Initiation of statin therapy within the last 12 weeks Lifestyle
* More than 10% weight loss or gain during the past 6 months
* Recent initiation (past 4 weeks) of exercise program
* Plan to become pregnant in the next 6 months
* Pregnancy or lactation
* Recent initiation or cessation of hormonal birth control or change in hormonal birth control regimen within the last 12 weeks
* Use of tobacco products
* More than 2 standard alcoholic drinks per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-06-17 (Actual); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Plasma inflammatory mediators | Change from 0 hour up to 6 hours postprandial
  Plasma cytokines will be measured using a multi-plex immunoassay and plasma oxylipins will be measured by mass spectroscopy.

SECONDARY OUTCOMES:
Plasma lipid profile | Change from 0 hour up to 6 hours postprandial
  Plasma lipids (triglycerides, total cholesterol, LDL-C, HDL-C) will be measured by enzymatic analysis by UC Davis Pathology Lab.
Plasma bone markers | Change from 0 hour up to 6 hours postprandial
  Plasma N-terminal telopeptide (NTX), C-terminal telopeptide (CTX) and propeptide of type I collagen (P1NP) will be measured by multi-plex immunoassay.
Urinary metabolites | Change from 0 hour up to 6 hours postprandial
  Urinary metabolites will be measured by nuclear magnetic resonance (NMR) spectroscopy.
Plasma glucose | Change from 0 hour up to 6 hours postprandial
  Plasma glucose will be measured by enzymatic analysis by UC Davis Pathology Lab.
Red blood cell functionality | Change from 0 hour up to 6 hours postprandial
  Red blood cells isolated from whole blood will be measured for sheer stress using an in-vitro microfluidic assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer T Smilowitz, PhD, Principal Investigator — UC Davis; Angela M. Zivkovic, PhD, Principal Investigator — University of California, Davis; Marta Van Loan, PhD, Principal Investigator — ARS USDA WHNRC; J. Bruce German, PhD, Principal Investigator — UC Davis; Bruce Hammock, PhD, Principal Investigator — UC Davis
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Background] Astrup A, Dyerberg J, Elwood P, Hermansen K, Hu FB, Jakobsen MU, Kok FJ, Krauss RM, Lecerf JM, LeGrand P, Nestel P, Riserus U, Sanders T, Sinclair A, Stender S, Tholstrup T, Willett WC. The role of reducing intakes of saturated fat in the prevention of cardiovascular disease: where does the evidence stand in 2010? Am J Clin Nutr. 2011 Apr;93(4):684-8. doi: 10.3945/ajcn.110.004622. Epub 2011 Jan 26. PMID 21270379
- [Background] Kratz M, Baars T, Guyenet S. The relationship between high-fat dairy consumption and obesity, cardiovascular, and metabolic disease. Eur J Nutr. 2013 Feb;52(1):1-24. doi: 10.1007/s00394-012-0418-1. Epub 2012 Jul 19. PMID 22810464
- [Background] Snow DR, Ward RE, Olsen A, Jimenez-Flores R, Hintze KJ. Membrane-rich milk fat diet provides protection against gastrointestinal leakiness in mice treated with lipopolysaccharide. J Dairy Sci. 2011 May;94(5):2201-12. doi: 10.3168/jds.2010-3886. PMID 21524510
- [Background] Dalbeth N, Gracey E, Pool B, Callon K, McQueen FM, Cornish J, MacGibbon A, Palmano K. Identification of dairy fractions with anti-inflammatory properties in models of acute gout. Ann Rheum Dis. 2010 Apr;69(4):766-9. doi: 10.1136/ard.2009.113290. Epub 2009 Aug 26. PMID 19713204
- [Background] Dalbeth N, Palmano K. Effects of dairy intake on hyperuricemia and gout. Curr Rheumatol Rep. 2011 Apr;13(2):132-7. doi: 10.1007/s11926-010-0160-8. PMID 21188562
- [Background] El Alwani M, Wu BX, Obeid LM, Hannun YA. Bioactive sphingolipids in the modulation of the inflammatory response. Pharmacol Ther. 2006 Oct;112(1):171-83. doi: 10.1016/j.pharmthera.2006.04.004. Epub 2006 Jun 8. PMID 16759708
- [Background] Dial EJ, Zayat M, Lopez-Storey M, Tran D, Lichtenberger L. Oral phosphatidylcholine preserves the gastrointestinal mucosal barrier during LPS-induced inflammation. Shock. 2008 Dec;30(6):729-33. doi: 10.1097/SHK.0b013e318173e8d4. PMID 18496240
- [Background] Park EJ, Suh M, Thomson B, Ma DW, Ramanujam K, Thomson AB, Clandinin MT. Dietary ganglioside inhibits acute inflammatory signals in intestinal mucosa and blood induced by systemic inflammation of Escherichia coli lipopolysaccharide. Shock. 2007 Jul;28(1):112-7. doi: 10.1097/SHK.0b013e3180310fec. PMID 17510604
- [Result] Beals E, Kamita SG, Sacchi R, Demmer E, Rivera N, Rogers-Soeder TS, Gertz ER, Van Loan MD, German JB, Hammock BD, Smilowitz JT, Zivkovic AM. Addition of milk fat globule membrane-enriched supplement to a high-fat meal attenuates insulin secretion and induction of soluble epoxide hydrolase gene expression in the postprandial state in overweight and obese subjects. J Nutr Sci. 2019 Apr 26;8:e16. doi: 10.1017/jns.2019.11. eCollection 2019. PMID 31080589
- [Result] Rogers TS, Demmer E, Rivera N, Gertz ER, German JB, Smilowitz JT, Zivkovic AM, Van Loan MD. The role of a dairy fraction rich in milk fat globule membrane in the suppression of postprandial inflammatory markers and bone turnover in obese and overweight adults: an exploratory study. Nutr Metab (Lond). 2017 May 17;14:36. doi: 10.1186/s12986-017-0189-z. eCollection 2017. PMID 28529534
- [Result] Demmer E, Van Loan MD, Rivera N, Rogers TS, Gertz ER, German JB, Smilowitz JT, Zivkovic AM. Addition of a dairy fraction rich in milk fat globule membrane to a high-saturated fat meal reduces the postprandial insulinaemic and inflammatory response in overweight and obese adults. J Nutr Sci. 2016 Mar 7;5:e14. doi: 10.1017/jns.2015.42. eCollection 2016. PMID 27313850